CLINICAL TRIAL: NCT02195427
Title: A Controlled, Randomized, Double-Blinded, Within-Subject, Multicenter, Prospective Clinical Study of TEOSYAL® RHA Global Action and TEOSYAL® RHA Deep Lines Versus Juvéderm® Ultra XC in the Treatment of Moderate to Severe Nasolabial Folds
Brief Title: TEOSYAL® RHA Global Action, TEOSYAL® RHA Deep Lines, and Juvéderm® Ultra XC for the Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEO-RHA-1302
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Nasolabial Folds, Wrinkles
Keywords: Nasolabial folds; Dermal filler; Hyaluronic acid (HA); Wrinkles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEOSYAL RHA Global Action/Juvederm Ultra XC (Experimental): Split-face injection of TEOSYAL® RHA Global Action into one NLF and Juvederm® Ultra XC into the contralateral NLF (n=75). Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  Interventions: Device: TEOSYAL® RHA Global Action
- TEOSYAL RHA Deep Lines/Juvederm Ultra XC (Experimental): Split-face injection of TEOSYAL® RHA Deep Lines into one NLF and Juvederm® Ultra XC into the contralateral NLF (n=75). Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  Interventions: Device: TEOSYAL® RHA Deep Lines

INTERVENTIONS:
Device: TEOSYAL® RHA Global Action — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 30G1/2" disposable sterile needles.
  Arms: TEOSYAL RHA Global Action/Juvederm Ultra XC
Device: TEOSYAL® RHA Deep Lines — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 27G1/2" disposable sterile needles.
  Arms: TEOSYAL RHA Deep Lines/Juvederm Ultra XC

SUMMARY:
The purpose of this study is 1) to compare the effectiveness and safety of TEOSYAL® RHA Global Action versus Juvéderm® Ultra XC, and 2) to compare the effectiveness and safety of TEOSYAL® RHA Deep Lines versus Juvéderm® Ultra XC, in the treatment of moderate to severe nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 22 years of age or older; female subjects of childbearing potential must have a negative urine pregnancy test and practice a reliable method of contraception
* NLFs classified as WSRS grade 3 or 4 (same score for each side)
* Willing to abstain from facial aesthetic procedures/therapies that could interfere with study evaluations
* Able to follow study instructions and likely to complete all required visits;
* Signed informed consent and HIPAA (Health Insurance Portability and Accountability Act) form

Exclusion Criteria:

* Female subjects that are pregnant or breast-feeding, or of childbearing potential and not practicing reliable birth control
* Known hypersensitivity/allergy to any component of the study devices
* Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, history of anaphylactic shock
* Known susceptibility to keloid formation, hypertrophic scarring or clinically significant skin pigmentation disorders
* Clinically significant active skin disease within 6 months
* History of active chronic debilitating systemic disease
* History of connective tissue disease
* History of malignancy (excl. non-melanoma skin cancer) within past 5 years
* History of bleeding disorders
* Need for clinically significant and continuous medical treatment within 2 weeks prior to first visit
* Received/used a prohibited treatment/procedure within certain time periods (e.g., bioresorbable fillers, NSAIDS, acetylsalicylic acid, high dose vitamin E, corticosteroids, interferon, anti-coagulation therapies, laser/light therapies, botulinum toxin injections (frontalis and glabella complex treatment permitted), prescription strength topical retinoids, facial peels, excisional facial surgery, clinically significant oral or maxillofacial surgery)
* Clinically significant alcohol or drug abuse, or history of poor cooperation, non-compliance with medical treatment, or unreliability
* Exhibit a physical attribute(s) that may prevent assessment or treatment of NLFs such as excessive facial hair, traumatic or surgical facial scars, and/or excessive hyperpigmentation in the treatment areas
* A condition or situation that may put the subject at significant risk, confound the study results, or significantly interfere with the subject participation

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - United States, Alabama, Birmingham, Alabama
  - United States, California, Beverly Hills, California
  - United States, Santa Monica, Santa Monica, California
  - United States, Florida, Coral Gables, Florida
  - United States, Massachusetts, Chestnut Hill, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 148 subjects were randomized to RHA Global Action (GA)/Juvederm (J) (n=74), RHA Deep Lines (DL)/Juvederm (J) (n=74).
  26 subjects were randomized to an untreated group (recruited only to avoid Blinded Live Evaluator to be biased so, not presented)
Pre-assignment Details: One subject randomized to the RHA GA/J withdrew consent prior to receiving initial treatment reducing the population for this cohort to n=73.
Groups:
- TEOSYAL RHA Global Action/Juvederm Ultra XC: Split-face injection of TEOSYAL® RHA Global Action into one NLF and Juvederm® Ultra XC into the contralateral NLF. Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  TEOSYAL® RHA Global Action: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 30G1/2" disposable sterile needles.
- TEOSYAL RHA Deep Lines/Juvederm Ultra XC: Split-face injection of TEOSYAL® RHA Deep Lines into one NLF and Juvederm® Ultra XC into the contralateral NLF. Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
  TEOSYAL® RHA Deep Lines: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus equi bacteria, formulated to a concentration of 23 mg/mL and 0.3% w/w lidocaine in a physiologic buffer. It is supplied in individual treatment syringes with 27G1/2" disposable sterile needles.
Period: Overall Study
Arm/Group | TEOSYAL RHA Global Action/Juvederm Ultra XC | TEOSYAL RHA Deep Lines/Juvederm Ultra XC
Started | 73 | 74
N Patients at W24 (Primary Outcome) | 67 | 62
N Patients at W36 | 65 | 59
N Patients at W52 | 63 | 56
Completed (N patients completed W64) | 47 | 47
Not Completed | 26 | 27
Not completed — Did not consent to study extension | 13 | 9
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 7 | 14
Not completed — Conditional re-treatment at W52 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- TEOSYAL RHA Global Action/Juvederm Ultra XC: Split-face injection of TEOSYAL® RHA Global Action into one NLF and Juvederm® Ultra XC into the contralateral NLF. Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
- TEOSYAL RHA Deep Lines/Juvederm Ultra XC: Split-face injection of TEOSYAL® RHA Deep Lines into one NLF and Juvederm® Ultra XC into the contralateral NLF. Up to 3.0 mL injected per NLF (mid-dermis to deep-dermis). Touch-up treatment provided at 2 weeks (up to 3.0 mL per NLF).
- Total: Total of all reporting groups
Arm/Group | TEOSYAL RHA Global Action/Juvederm Ultra XC | TEOSYAL RHA Deep Lines/Juvederm Ultra XC | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.9) | 55.7 (9.4) | 55.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 68 | 130
  Male | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 59 | 62 | 121
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 74 | 147
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color.
  Type I - always burns, never tans (pale white; blond or red hair; blue eyes; freckles).
  Type II - usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes) Type III - sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV - burns minimally, always tans well (moderate brown) Type V - very rarely burns, tans very easily (dark brown) Type VI - Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Types I to III | 45 | 44 | 89
    Types IV to VI | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of the Delta of TEOSYAL® RHA GA and TEOSYAL® RHA DL Versus Juvéderm® Ultra XC for the Correction of Moderate to Severe NLFs Based on the Wrinkle Severity Rating Scale (WSRS) Score Assessed by the Blinded Live Evaluator (BLE).
Description: TEOSYAL® RHA GA = TEOSYAL® RHA Global Action TEOSYAL® RHA DL = TEOSYAL® RHA Deep Lines WSRS (Wrinkle Severity Rating Scale) is a validated 5-point scale assessing wrinkle severity with 1 being 'absent' and 5 being 'extreme' BLE = Blinded Live Evaluator
Time Frame: Baseline and 24 weeks after last treatment
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Groups:
- TEOSYAL® RHA Global Action: Injection of TEOSYAL® RHA Global Action into one NLF
- Juvéderm® Ultra XC (RHA GA): Injection of Juvéderm® Ultra XC into the contralateral NLF of the one injected with TEOSYAL® RHA Global Action
- TEOSYAL® RHA Deep Lines: Injection of TEOSYAL® RHA Deep Lines into one NLF
- Juvéderm® Ultra XC (RHA DL): Injection of Juvéderm® Ultra XC into the contralateral NLF of the one injected with TEOSYAL® RHA Deep Lines
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
units on a scale | -1.16 [-1.36 to -0.97] | -1.13 [-1.33 to -0.93] | -1.32 [-1.53 to -1.12] | -1.23 [-1.43 to -1.02]
Statistical Analysis 1: Comparison: TEOSYAL® RHA Global Action vs Juvéderm® Ultra XC (RHA GA); Efficacy of TEOSYAL® RHA Global Action versus control is analyzed in a non-inferiority statistical model using the 5-grade Wrinkle Severity Rating Scale (WSRS) as rated by the Blinded Live Evaluator at 24 weeks after baseline. The primary endpoint is the aesthetic improvement from pre-injection of the NLF at the side of the face treated with TEOSYAL® RHA Ultra Deep compared to the one at the side of the face treated with the control device, as assessed by the BLE at 24 weeks after baseline; Test type: Non-Inferiority — A WSRS change of 1 grade is considered to be clinically significant. A difference of ≤0.5 grade between the two treatment groups (i.e., half of the clinically significant difference) = non-inferiority margin. The primary efficacy endpoint uses a paired-design and is analyzed by calculating two-sided confidence intervals of the mean difference between TEOSYAL® RHA Global Action and the control device, between the V1 enrollment visit (baseline) and V7 (24 weeks after baseline); Mean Difference (Final Values) = -0.03, 97.5% CI 2-sided [-0.17 to 0.11] — The decision is based on the upper limit of the 2-sided confidence interval for the difference for the change from baseline, between test and comparator treatment. For achieving non-inferiority, the upper confidence limit of a 97.5% CI must be ≤0.5
Statistical Analysis 2: Comparison: TEOSYAL® RHA Deep Lines vs Juvéderm® Ultra XC (RHA DL); Efficacy of TEOSYAL® RHA Deep Lines versus control is analyzed in a non-inferiority statistical model using the 5-grade Wrinkle Severity Rating Scale (WSRS) as rated by the Blinded Live Evaluator at 24 weeks after baseline. The primary endpoint is the aesthetic improvement from pre-injection of the NLF at the side of the face treated with TEOSYAL® RHA Deep Lines compared to the one at the side of the face treated with the control device, as assessed by the BLE at 24 weeks after baseline; Test type: Non-Inferiority — A WSRS change of 1 grade is considered to be clinically significant. A difference of ≤0.5 grade between the two treatment groups (i.e., half of the clinically significant difference) = non-inferiority margin. The primary efficacy endpoint uses a paired-design and is analyzed by calculating two-sided confidence intervals of the mean difference between TEOSYAL® RHA Deep Lines and the control device, between the V1 enrollment visit (baseline) and V7 (24 weeks after baseline); Mean Difference (Final Values) = -0.10, 97.5% CI 2-sided [-0.25 to 0.06] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Post Injection Treatment Responses (From Common Treatment Responses (CTR) Diary) for Safety Evaluation of TEOSYAL® RHA Global Action (GA) and TEOSYAL® RHA Deep Lines (DL) Versus Juvéderm® Ultra XC (J).
Description: The subjects received a diary booklet and instructions for recording his/her observations of the Common Treatment Responses of the study treatments for the first 14 days after each treatment (initial, touch-up). The diary was discussed during each telephone follow-up visit. Subjects should complete the diary at approximately the same time each day (i.e., am or pm).
  The subject diary captured the following Common Treatment Responses (CTR) that occur following the injection of a dermal filler; specifically, redness, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching, discoloration, and "other".
  The 14-day patient CTR diary included a detailed glossary describing all signs/symptoms listed in the diary; an option was provided to rate "other" if the subject experienced a sign/symptom that is not listed.
  The table presents the number of subjects experiencing at least 1 Common Treatment Response (CTR)
Time Frame: During 14 days after initial treatment (D0) and touch-up (2 weeks)
Population: 1 subject randomized to the GA/J cohort received injections with DL/J and was placed in the DL/J cohort for safety evaluation; So: N=75 for DL/J SAFT population and N=72 for GA/J SAFT population.
  Number of patients for CTR after touch-up treatment are based on number of patients receiving Touch-up treatment (GA N=47/J-GA N=49/DL N=50/J-DL N=53)
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 72 | 72 | 75 | 75
Participants
  Bruising (initial treatment) | 36 | 41 | 42 | 38
  Bruising (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Bruising (Touch-up) | 15 | 13 | 19 | 20
  Discolouration (initial treatment) | 24 | 27 | 22 | 22
  Discolouration (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Discolouration (Touch-up) | 11 | 13 | 10 | 12
  Firmness (initial treatment) | 46 | 48 | 48 | 45
  Firmness (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Firmness (Touch-up) | 25 | 20 | 34 | 31
  Itching (initial treatment) | 12 | 15 | 13 | 11
  Itching (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Itching (Touch-up) | 5 | 4 | 5 | 5
  Lumps/Bumps (initial treatment) | 38 | 37 | 49 | 40
  Lumps/Bumps (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Lumps/Bumps (Touch-up) | 21 | 17 | 30 | 24
  Pain (initial treatment) | 19 | 16 | 30 | 23
  Pain (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Pain (Touch-up) | 10 | 9 | 16 | 19
  Redness (initial treatment) | 45 | 49 | 43 | 42
  Redness (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Redness (Touch-up) | 15 | 16 | 27 | 25
  Swelling (initial treatment) | 42 | 45 | 41 | 38
  Swelling (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Swelling (Touch-up) | 23 | 22 | 31 | 31
  Tenderness (Initial treatment) | 44 | 40 | 44 | 37
  Tenderness (Touch-up): number analyzed (Participants) | 47 | 49 | 50 | 53
  Tenderness (Touch-up) | 22 | 18 | 29 | 27

3. Secondary Outcome: Assessment of Injection Site Pain (Visual Analog Scale) of TEOSYAL® RHA Global Action (GA) and TEOSYAL® RHA Deep Lines (DL) Versus Juvéderm® Ultra XC (J).
Description: VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain
Time Frame: During Injection and 5, 15, 30 minutes post-injection
Population: 1 subject randomized to the GA/J cohort received injections with DL/J and was placed in the DL/J cohort for safety evaluation; So: N=75 for DL/J SAFT population and N=72 for GA/J SAFT population.
  Number of patients after touch-up treatment are based on number of patients receiving Touch-up treatment (GA N=47/J-GA N=49/DL N=50/J-DL N=53)
Measure: Mean (Standard Deviation); unit: VAS score
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 72 | 72 | 75 | 75
VAS score
  Initial injection mean pain during injection | 15.0 (17.2) | 13.9 (17.4) | 16.7 (17.8) | 14.6 (17.7)
  Initial injection mean pain 5 min post-injection | 3.8 (9.1) | 3.9 (9.5) | 3.7 (7.7) | 2.9 (5.1)
  Initial injection mean pain 15 min post-injection | 1.1 (3.3) | 1.4 (3.9) | 2.0 (5.5) | 1.4 (3.2)
  Initial injection mean pain 30 min post-injection | 0.5 (1.7) | 0.7 (1.9) | 1.0 (3.0) | 0.5 (0.9)
  Touch-up injection mean pain during injection: number analyzed (Participants) | 47 | 49 | 50 | 53
  Touch-up injection mean pain during injection | 12.6 (17.5) | 11.8 (14.6) | 15.9 (17.4) | 14.5 (18.4)
  Touch-up injection mean pain 5 min post-injection: number analyzed (Participants) | 47 | 49 | 50 | 53
  Touch-up injection mean pain 5 min post-injection | 3.2 (9.1) | 2.8 (7.3) | 4.6 (9.7) | 3.5 (7.3)
  Touch-up injection mean pain 15 min post-injection: number analyzed (Participants) | 47 | 49 | 50 | 53
  Touch-up injection mean pain 15 min post-injection | 1.7 (7.1) | 1.3 (5.8) | 2.2 (5.2) | 1.9 (4.6)
  Touch-up injection mean pain 30 min post-injection: number analyzed (Participants) | 47 | 49 | 50 | 53
  Touch-up injection mean pain 30 min post-injection | 1.2 (5.2) | 1.0 (5.0) | 1.5 (4.6) | 1.2 (3.9)

4. Secondary Outcome: Delta of the WSRS Score Between W24,36,52 and Baseline for TEOSYAL® RHA GA Versus Juvéderm® Ultra XC and TEOSYAL® RHA DL Versus Juvéderm® Ultra XC for the Correction of Moderate to Severe NLFs Based on the WSRS Score Assessed by the BLE
Description: as for outcome 1
Time Frame: Baseline and Weeks 24, 36, 52, 64
Population: Numbers of patients analyzed correspond to patients that have completed the visits and for which data were available (See participant flow)
Measure: Mean (Standard Deviation); unit: WSRS Delta from V1
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
WSRS Delta from V1
  W24 Delta from V1 | -1.16 (0.69) | -1.13 (0.72) | -1.32 (0.70) | -1.23 (0.71)
  W36 Delta from V1: number analyzed (Participants) | 65 | 65 | 58 | 58
  W36 Delta from V1 | -1.12 (0.65) | -1.12 (0.60) | -1.03 (0.70) | -0.98 (0.69)
  W52 Delta from V1: number analyzed (Participants) | 62 | 62 | 56 | 56
  W52 Delta from V1 | -1.06 (0.60) | -1.06 (0.65) | -0.91 (0.77) | -0.82 (0.74)
  W64 Delta fom V1: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 Delta fom V1 | -0.94 (0.57) | -1.00 (0.63) | -0.91 (0.72) | -0.83 (0.67)

5. Secondary Outcome: Delta of the WSRS Score Between W2,4,12,24,36,52,64 and Baseline for TEOSYAL® RHA GA Versus Juvéderm® Ultra XC and TEOSYAL® RHA Deep Lines Versus Juvéderm® Ultra XC for the Correction of Moderate to Severe NLFs Based on the WSRS Score Assessed by the TI
Description: TEOSYAL® RHA GA = TEOSYAL® RHA Global Action TEOSYAL® RHA DL = TEOSYAL® RHA Deep Lines WSRS (Wrinkle Severity Rating Scale) is a validated 5-point scale assessing wrinkle severity with 1 being 'absent' and 5 being 'extreme' TI = Treating Investigator
Time Frame: Baseline and Weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: WSRS Delta from V1
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
WSRS Delta from V1
  W2 Delta from V1 | -1.49 (0.61) | -1.34 (0.73) | -1.45 (0.64) | -1.31 (0.59)
  W4 Delta from V1: number analyzed (Participants) | 65 | 65 | 61 | 61
  W4 Delta from V1 | -1.66 (0.64) | -1.69 (0.64) | -1.84 (0.45) | -1.77 (0.50)
  W12 Delta from V1: number analyzed (Participants) | 65 | 65 | 62 | 62
  W12 Delta from V1 | -1.52 (0.69) | -1.32 (0.77) | -1.65 (0.55) | -1.58 (0.56)
  W24 Delta from V1 | -1.33 (0.59) | -1.25 (0.70) | -1.55 (0.59) | -1.39 (0.55)
  W36 Delta from V1: number analyzed (Participants) | 65 | 65 | 59 | 59
  W36 Delta from V1 | -1.23 (0.61) | -1.17 (0.72) | -1.08 (0.65) | -1.03 (0.67)
  W52 Delta from V1: number analyzed (Participants) | 63 | 63 | 56 | 56
  W52 Delta from V1 | -1.24 (0.64) | -1.16 (0.63) | -1.07 (0.68) | -0.93 (0.57)
  W64 Delta from V1: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 Delta from V1 | -1.09 (0.58) | -0.98 (0.61) | -0.98 (0.57) | -0.89 (0.63)

6. Secondary Outcome: Percentage of Responders Based on the Intra-individual Improvement of at Least One Grade in the WSRS Compared to Baseline Assessed by the BLE
Description: A responder correspond to a subject with an intra-individual improvement of at least one grade in the WSRS compared to baseline
Time Frame: Baseline and Weeks 24, 36, 52, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
percentage of responders
  W24 | 83.6 [72.5 to 91.5] | 82.1 [70.8 to 90.4] | 91.9 [82.2 to 97.3] | 88.7 [78.1 to 95.3]
  W36: number analyzed (Participants) | 65 | 65 | 58 | 58
  W36 | 86.2 [75.3 to 93.5] | 87.7 [77.2 to 94.5] | 82.8 [70.6 to 91.4] | 79.3 [66.7 to 88.8]
  W52: number analyzed (Participants) | 62 | 62 | 56 | 56
  W52 | 85.5 [74.2 to 93.1] | 82.3 [70.5 to 90.8] | 75.0 [61.6 to 85.6] | 69.6 [55.9 to 81.2]
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 80.9 [66.7 to 90.6] | 80.9 [66.7 to 90.9] | 78.7 [64.3 to 89.3] | 72.3 [57.4 to 84.4]

7. Secondary Outcome: Percentage of Responders Based on the Intra-individual Improvement of at Least One Grade in the WSRS Compared to Baseline Assessed by the TI
Description: as for outcome 6
Time Frame: Baseline and Weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
percentage of responders
  W2 | 98.5 [92.0 to 100.0] | 91.0 [81.5 to 96.6] | 95.2 [86.5 to 99.0] | 93.6 [84.3 to 98.2]
  W4: number analyzed (Participants) | 65 | 65 | 61 | 61
  W4 | 98.5 [91.7 to 100.0] | 98.5 [91.7 to 100.0] | 100.0 [94.1 to 100.0] | 100.0 [94.1 to 100.0]
  W12: number analyzed (Participants) | 65 | 65 | 62 | 62
  W12 | 95.4 [87.1 to 99.0] | 87.7 [77.2 to 94.5] | 100.0 [94.2 to 100.0] | 100.0 [94.2 to 100.0]
  W24 | 94.0 [85.4 to 98.4] | 86.6 [76.0 to 93.7] | 96.8 [88.8 to 99.6] | 98.4 [91.3 to 100.0]
  W36: number analyzed (Participants) | 65 | 65 | 59 | 59
  W36 | 90.8 [81.0 to 96.5] | 83.1 [71.7 to 91.2] | 83.1 [71.0 to 91.6] | 79.7 [67.2 to 89.0]
  W52: number analyzed (Participants) | 63 | 63 | 56 | 56
  W52 | 88.9 [78.4 to 95.4] | 87.3 [76.5 to 94.4] | 80.4 [67.6 to 89.8] | 80.4 [67.6 to 89.8]
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 87.2 [74.3 to 95.2] | 80.9 [66.7 to 90.0] | 83.0 [69.2 to 92.4] | 74.5 [59.7 to 86.1]

8. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) Scale by the Blinded Live Evaluator (BLE).
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse" that evaluate the aesthetic improvement from baseline.
  GAI was assessed using the baseline photograph. Each side of the face was assessed independently.
Time Frame: Weeks 24, 36, 52, 64
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
Participants
  W24: number analyzed (Participants) | 67 | 67 | 61 | 61
  W24 | 61 | 59 | 59 | 58
  W36: number analyzed (Participants) | 65 | 65 | 58 | 58
  W36 | 60 | 61 | 53 | 50
  W52: number analyzed (Participants) | 62 | 62 | 56 | 56
  W52 | 57 | 54 | 46 | 44
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 41 | 39 | 40 | 37

9. Secondary Outcome: Number of Global Aesthetic Improvement (GAI) Responders (i.e., Scoring Either "Much Improved" or "Improved") on GAI Scale.
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse" that evaluate the aesthetic improvement from baseline.
  GAI was assessed using the baseline photograph. Subjects will be instructed: "Use a mirror to compare your face to the photograph provided to you and rate the degree of aesthetic improvement by using the following scale".
  Each side of the face was assessed independently.
Time Frame: Weeks 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
Participants
  W4: number analyzed (Participants) | 65 | 65 | 61 | 61
  W4 | 64 | 63 | 59 | 59
  W12: number analyzed (Participants) | 65 | 65 | 62 | 62
  W12 | 60 | 59 | 59 | 60
  W24 | 59 | 59 | 55 | 55
  W36: number analyzed (Participants) | 65 | 65 | 59 | 59
  W36 | 59 | 58 | 54 | 53
  W52: number analyzed (Participants) | 62 | 62 | 56 | 56
  W52 | 55 | 53 | 50 | 49
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 44 | 45 | 43 | 41

10. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q (NLF Domain) Questionnaire
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  FACE-Q questionnaire is composed of 5 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  The subject was instructed as follows: "These questions ask about how you look right now. With your nasolabial folds in mind (the deep lines that run downward from the sides of your nose), in the past week, how much have you been bothered by:", and provided response.
  * How deep your nasolabial fold are?
  * How your nasolabial folds look when your face is relaxed (still)?
  * How old your nasolabial folds make you look?
  * How your nasolabial folds look when you smile?
  * How your nasolabial folds look compared with other people your age? To calculate the FACE-Q, outcomes from all 5 questions were pooled and adapted to a scale to 100 units. Data were also transformed so that higher scores reflected a beneficial outcome.
Time Frame: Immediately post-injection, and weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
units on a scale
  pre-treatment | 24.7 (17.7) | 25.2 (16.5) | 29.1 (17.0) | 27.7 (17.8)
  W2 | 70.3 (22.7) | 69.0 (22.2) | 67.4 (25.5) | 66.9 (25.3)
  W4: number analyzed (Participants) | 65 | 65 | 61 | 61
  W4 | 76.7 (22.1) | 75.6 (22.0) | 77.5 (20.4) | 78.0 (20.4)
  W12: number analyzed (Participants) | 65 | 65 | 62 | 62
  W12 | 74.5 (23.5) | 73.1 (23.7) | 77.5 (21.8) | 77.2 (21.9)
  W24 | 64.6 (24.8) | 62.9 (24.5) | 64.8 (24.5) | 66.2 (23.7)
  W36: number analyzed (Participants) | 65 | 65 | 59 | 59
  W36 | 64.0 (25.2) | 61.4 (25.1) | 66.0 (26.4) | 65.3 (25.2)
  W52: number analyzed (Participants) | 62 | 62 | 55 | 55
  W52 | 63.6 (29.3) | 61.8 (30.0) | 63.0 (27.4) | 60.5 (27.6)
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 58.4 (21.9) | 59.5 (22.4) | 64.1 (25.2) | 62.7 (24.9)

11. Secondary Outcome: Subject's Satisfaction Score
Description: Subjective 5-point scale with 1 being 'very satisfied' and 5 being 'very dissatisfied'
Time Frame: Weeks 2, 4, 12, 24, 36, 52, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
units on a scale
  W2 | 1.58 (0.72) | 1.57 (0.74) | 1.87 (0.78) | 1.81 (0.70)
  W4: number analyzed (Participants) | 65 | 65 | 61 | 61
  W4 | 1.29 (0.49) | 1.29 (0.49) | 1.43 (0.67) | 1.34 (0.54)
  W12: number analyzed (Participants) | 65 | 65 | 62 | 62
  W12 | 1.46 (0.64) | 1.55 (0.71) | 1.50 (0.76) | 1.50 (0.70)
  W24 | 1.73 (0.73) | 1.75 (0.75) | 1.63 (0.83) | 1.55 (0.74)
  W36: number analyzed (Participants) | 65 | 65 | 59 | 59
  W36 | 1.66 (0.76) | 1.69 (0.75) | 1.56 (0.82) | 1.63 (0.83)
  W52: number analyzed (Participants) | 62 | 62 | 56 | 56
  W52 | 1.47 (0.69) | 1.58 (0.78) | 1.55 (0.93) | 1.66 (0.82)
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 1.68 (0.75) | 1.66 (0.70) | 1.36 (0.67) | 1.45 (0.75)

12. Secondary Outcome: Volume to Obtain Optimal Cosmetic Result (Initial Treatment + Touch-up)
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
mL | 1.54 (0.66) | 1.30 (0.53) | 1.52 (0.62) | 1.30 (0.55)

13. Secondary Outcome: Number of Subjects Receiving Touch-up Treatment.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
Participants | 43 | 45 | 45 | 47

14. Secondary Outcome: Number of Subjects Receiving Re-treatment
Time Frame: Weeks 24, 36, 52, 64
Population: Numbers of patients analyzed correspond to patients that have completed the visits (See participant flow)
Measure: Count of Participants; unit: Participants
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Number analyzed (Participants) | 67 | 67 | 62 | 62
Participants
  W24 | 1 | 1 | 0 | 0
  W36: number analyzed (Participants) | 65 | 65 | 59 | 59
  W36 | 3 | 3 | 5 | 5
  W52: number analyzed (Participants) | 63 | 63 | 56 | 56
  W52 | 9 | 11 | 9 | 9
  W64: number analyzed (Participants) | 47 | 47 | 47 | 47
  W64 | 42 | 43 | 39 | 38

ADVERSE EVENTS:
Time Frame: 64 weeks or 68 weeks for patients receiving a re-treatment at W64
Description: The TI assessed all AEs and recorded details of seriousness, severity, duration, and action taken with study device, and relationship to the study device.
  1 subject randomized to the RHA Global Action/Juverderm cohort received injections with RHA Deep Lines/Juvederm and was placed in the RHA Deep Lines/Juvederm cohort for safety evaluation; So: N=75 for RHA Deep Lines/Juvederm SAFT population and N=72 for RHA Global Action/Juvederm SAFT population.
Arm/Group | TEOSYAL® RHA Global Action | Juvéderm® Ultra XC (RHA GA) | TEOSYAL® RHA Deep Lines | Juvéderm® Ultra XC (RHA DL)
Serious Adverse Events (participants affected / at risk) | 2/75 | 2/75 | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 39/72 | 36/72 | 30/75 | 31/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEOSYAL® RHA Global Action (N=75) | Juvéderm® Ultra XC (RHA GA) (N=75) | TEOSYAL® RHA Deep Lines (N=75) | Juvéderm® Ultra XC (RHA DL) (N=75)
Gastric Ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — unrelated to the study device
Gatric Ulcer Perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — unrelated to the study device
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEOSYAL® RHA Global Action (N=72) | Juvéderm® Ultra XC (RHA GA) (N=72) | TEOSYAL® RHA Deep Lines (N=75) | Juvéderm® Ultra XC (RHA DL) (N=75)
Injection site firmness (General disorders) | 20 (25) | 17 (20) | 19 (25) | 9 (12)
Injection site lumps/bumps (General disorders) | 15 (18) | 7 (9) | 17 (22) | 14 (16)
Injection site haematoma (General disorders) | 5 (6) | 4 (5) | 5 (6) | 5 (6)
Tenderness (General disorders) | 7 (8) | 3 (3) | 10 (11) | 4 (4)
Injection site discolouration (General disorders) | 3 (3) | 5 (5) | 4 (4) | 4 (4)
Injection site pain (General disorders) | 4 (4) | 4 (4) | 2 (2) | 2 (2)
Injection site swelling (General disorders) | 6 (7) | 3 (4) | 9 (11) | 5 (7)
Injection site erythema (General disorders) | 2 (2) | 4 (4) | 5 (7) | 5 (7)
Injection site pruritus (General disorders) | 4 (5) | 3 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days